CLINICAL TRIAL: NCT02696538
Title: Comparative Utility of the Mini-BESTest, Berg Balance Scale, and Functional Gait Assessment to Predict Falls in Individuals After Traumatic Brain Injury
Brief Title: Comparative Utility of Clinical Balance Measures in Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Marissa Lyon, Physical Therapist, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC-MH-15-0656
Record Dates: First submitted 2016-02-26; First posted 2016-03-02 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Traumatic Brain Injury; Acquired Brain Injury; Accidental Falls
Keywords: Fall risk; Rehabiliation; Physical Therapy; Functional Gait Assessment; mini-Balance Evaluation Systems Test; Berg Balance Scale; Psychometric properties; Validity; Inter-rater reliability; Montreal Cognitive Assessment
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): All participants included in this group and will complete all three outcomes assessment
  Interventions: Other: Functional Gait Assessment; Other: mini-Balance Evaluation Systems Test; Other: Berg Balance Scale

INTERVENTIONS:
Other: Functional Gait Assessment — Balance assessment
Other: mini-Balance Evaluation Systems Test — Balance assessment
Other: Berg Balance Scale — Balance assessment

SUMMARY:
The purpose of this research study is to investigate how useful three balance tests are in predicting fall risk in the individual with traumatic brain injury (TBI). These tests are the Functional Gait Assessment (FGA), the Berg Balance Scale (BBS), and the mini-Balance Evaluation Systems Test (mini-BESTest).

DETAILED DESCRIPTION:
The purpose of the proposed study is to investigate the reliability and predictive validity of three balance measures, the Berg Balance Scale (BBS), the Functional Gait Assessment (FGA) and the mini-Balance Evaluation Systems Test (mini-BESTest), among individuals with history of traumatic brain injury. Participants will complete a health history questionnaire and six-month fall history. When available, fall history will be corroborated with a family member that resides with the participant. Participants will complete the Montreal Cognitive Assessment. Each participant will then participate in a 45-minute evaluation using the three performance-based outcome measures, with order randomized, with two blinded assessors. Six and 12 month follow-up of number of falls will occur via telephone. Statistical analysis with investigate the inter-rater reliability, predictive validity of fall risk and to determine cut off scores for fallers vs. non fallers in the population.

ELIGIBILITY:
Inclusion Criteria:

* community dwelling
* medically stable
* able to stand at least one minute unsupported (with/without assistive device)
* able to ambulate 20 feet (with/without assistance or assistive device)
* able to follow one step instructions or visual demonstrations.

Exclusion Criteria:

* presence of partial or non-weight bearing on a lower extremity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-11 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-02-16 (Actual)

PRIMARY OUTCOMES:
total score on Functional Gait Assessment | Baseline
total score on Berg Balance Scale | Baseline
total on mini-Balance Evaluation System Test | Baseline
reported fall history | six month
  a fall is defined as unplanned and unexpected contact with the floor or lower surface not due to medical emergency (stroke, seizure, cardiac event) or environmental hazards (chair collapsing, earthquake)
reported fall history | twelve month
  a fall is defined as unplanned and unexpected contact with the floor or lower surface not due to medical emergency (stroke, seizure, cardiac event) or environmental hazards (chair collapsing, earthquake)

SECONDARY OUTCOMES:
Montreal Cognitive Assessment | Baseline
  assessment of mild cognitive deficits

CONTACTS AND LOCATIONS:
Overall Officials: Marissa F Lyon, DPT, Principal Investigator — Memorial Hermann
Locations (1):
- Marissa Lyon, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No